CLINICAL TRIAL: NCT06749067
Title: The Effect Of Mındfulness-Based and Occupatıonal Practıces On Psychologıcal Well-Beıng and Menopausal Symptoms In Menopausal Women: A Randomısed Controlled Trıal
Brief Title: Effect Of Awareness and Occupatıonal Practıces On Menopausal Women's Psychologıcal Wellbeıng And Menopausal Symptoms
Acronym: Mindfulness
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafkas University (Other)
Responsible Party: Principal Investigator, Şafak AYDİN, ASSISTANT PROFESSOR, Kafkas University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KafkasÜ-safak-36
Record Dates: First submitted 2024-12-19; First posted 2024-12-27 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Mindfulness Meditation; Occupational Therapy; Psychological Well-Being; Menopause
Keywords: Mindfulness; Nurse; Menopause; Occupational Practices; Psychological Well-Being
MeSH Terms: conditions — Psychological Well-Being | interventions — Mindfulness; Occupational Therapy

STUDY DESIGN:
Intervention Model Description: Women will be divided into three experimental and one control group by lottery method from the selected family health centre. All participants will first be informed about the intervention application and informed consent will be obtained. Afterwards, all participants will be asked to fill out the Personal Information Form, Psychological Well-Being Scale, Menopause Symptoms Assessment Scale as a pre-test application.
  As an intervention programme, no treatment will be applied to the women in the control group, Mindfulness-Based Practices for the women in the experimental 1 group, Engagement Practice for the experimental 2 group, and Mindfulness-Based Occupational Practice for the experimental 3 group were planned as 2 sessions per week for 8 weeks and 16 sessions of 45-60 minutes.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experiment 1 Group: Mindfulness Based Practices (Experimental): Experiment 1 Group Intervention: In the first session preparation session; face-to-face meeting with the women in the experimental group and then general information about the definition, purpose and applications of the mindfulness-based practice will be given, and the lack of information about the practice, if any, will be eliminated by receiving feedback from the women. The importance of regular and timely participation in the application will be emphasised, application days will be determined and phone numbers will be taken to contact women for online applications. Then, the pre-test data consisting of Personal Information Form, Psychological Well-Being Scale, Menopause Symptoms Assessment Scale will be filled out by obtaining voluntary consent.
  Interventions: Behavioral: Mindfulness Based Practices
- Experiment 2 Group: Occupational Practices (Experimental): Experiment 2 Group Intervention: In the first session preparation session, the women in the experimental group will be introduced face-to-face and then general information will be given about the definition, purpose and applications of the occupational practice, and the lack of information about the practice will be eliminated by receiving feedback from the women. The importance of regular and timely participation in the application will be emphasised, application days will be determined and phone numbers will be taken to contact women for online applications. Then, the pre-test data consisting of Personal Information Form, Psychological Well-Being Scale, Menopause Symptoms Assessment Scale will be filled out by obtaining voluntary consent.
  Interventions: Behavioral: Occupational Practices
- Experiment 3 Group: Mindfulness-Based Occupational Practice (Experimental): Experiment 3 Group Intervention: In the first session preparation session, the women in the experimental group will be introduced face-to-face and then general information will be given about the definition, purpose and applications of the occupational practice, and the lack of information about the practice will be eliminated by receiving feedback from the women. The importance of regular and timely participation in the application will be emphasised, application days will be determined and phone numbers will be taken to contact women for online applications. Then, the pre-test data consisting of Personal Information Form, Psychological Well-Being Scale, Menopause Symptoms Assessment Scale will be filled out by obtaining voluntary consent.
  In the first session, before starting the Mindfulness-Based Engagement Practice, women will be focused on the moment with a 3-minute breathing exercise, followed by a raisin exercise.
  Interventions: Behavioral: Mindfulness-Based Occupational Practice
- Control Group (No Intervention): Control Group: Telephone numbers will be taken to communicate with menopausal women who meet the inclusion criteria for the study. Then, the pre-test data consisting of Personal Information Form, Psychological Well-Being Scale, Menopause Symptoms Assessment Scale will be filled out by obtaining voluntary consent. No treatment will be applied to women in this group. At the end of 8 weeks, all participants will be asked to complete the Personal Information Form, Psychological Well-Being Scale, Menopause Symptoms Assessment Scale as a post-test application.

INTERVENTIONS:
Behavioral: Mindfulness Based Practices — Experiment 1 Group Intervention: In the first session preparation session; face-to-face meeting with the women in the experimental group and then general information about the definition, purpose and applications of the mindfulness-based practice will be given, and the lack of information about the practice, if any, will be eliminated by receiving feedback from the women. The importance of regular and timely participation in the application will be emphasised, application days will be determined and phone numbers will be taken to contact women for online applications. Then, the pre-test data consisting of Personal Information Form, Psychological Well-Being Scale, Menopause Symptoms Assessment Scale will be filled out by obtaining voluntary consent. In the first session, before starting the Awareness Practice, women will be focused on the moment with a 3-minute breathing exercise and then continue with the raisin exercise.
  Other Names: Mindfulness
  Arms: Experiment 1 Group: Mindfulness Based Practices
Behavioral: Occupational Practices — Experiment 2 Group Intervention: In the first session preparation session, the women in the experimental group will be introduced face-to-face and then general information will be given about the definition, purpose and applications of the occupational practice, and the lack of information about the practice will be eliminated by receiving feedback from the women. The importance of regular and timely participation in the application will be emphasised, application days will be determined and phone numbers will be taken to contact women for online applications. Then, the pre-test data consisting of Personal Information Form, Psychological Well-Being Scale, Menopause Symptoms Assessment Scale will be filled out by obtaining voluntary consent. Before starting the Busyness Practice, women will be asked to choose the practice that they can do within the scope of the busyness practice such as 'hand knitting, wood painting, charcoal, origami, bead work, jewellery design, painting tables with
  Other Names: Occupational Therapy
  Arms: Experiment 2 Group: Occupational Practices
Behavioral: Mindfulness-Based Occupational Practice — Experiment 3 Group Intervention: In the first session preparation session, the women in the experimental group will be introduced face-to-face and then general information will be given about the definition, purpose and applications of the occupational practice, and the lack of information about the practice will be eliminated by receiving feedback from the women. The importance of regular and timely participation in the application will be emphasised, application days will be determined and phone numbers will be taken to contact women for online applications. Then, the pre-test data consisting of Personal Information Form, Psychological Well-Being Scale, Menopause Symptoms Assessment Scale will be filled out by obtaining voluntary consent. In the first session, before starting the Mindfulness-Based Engagement Practice, women will be focused on the moment with a 3-minute breathing exercise, followed by a raisin exercise.
  Other Names: Mindfulness-Based; Occupational Therapy
  Arms: Experiment 3 Group: Mindfulness-Based Occupational Practice

SUMMARY:
Non-drug methods are frequently preferred in menopausal symptoms, especially in mental effects, and their effectiveness on symptoms is remarkable. Non-drug methods mainly used in the management of postmenopausal symptoms are sports, avoiding bad habits, paying attention to diet and increasing fluid intake, wearing comfortable clothes. In addition, there are many supportive methods such as stress reduction meditation practices, garden therapies, breathing and physical exercise practices, aromatherapy. Among the most frequently used coping methods of women experiencing menopausal symptoms such as irritability and anxiety/anxiety, it was found that 'paying attention to different things (housework, cleaning, cooking, handicrafts, etc.)' was among the most frequently used coping methods. In this direction, it is thought that occupational practice may have positive effects on menopausal symptoms in women. Engagement practices are one of the methods widely used in recent years to cope with anxiety, depression and stress.

Our study aimed to measure the effectiveness of mindfulness-based practices on menopausal symptoms and psychological well-being in menopausal women by blending mindfulness-based practices and busyness practices, and in this sense, it is anticipated that it will make a significant contribution to the literature.

Objective: This study will be conducted to determine the effect of mindfulness-based and occupational practices on psychological well-being and menopausal symptoms in menopausal women.

Materials and Methods: The research will be conducted as a randomised controlled experimental study in a four-group, parallel, pretest-posttest design. The research is planned to be conducted between December 2024 and December 2025. The population of the study consists of women in menopause who applied to the ASM in the centre of Kars between December 2024 and December 2025. The sample of the study will consist of women who meet the inclusion criteria among these women. As a result of the power analysis performed in the G*Power version 3.1.9.7 programme, it was determined that a total of 76 participants, at least 19 people in each of the intervention and control groups, with a sample size, 95% confidence, 95% test power (1-ß), 0.05% margin of error level, d = 0.25 effect size (Kang, 2021). Considering 10% possible data loss in the study, it was planned to include 20 women in each of the intervention and control groups.

DETAILED DESCRIPTION:
The transition from the reproductive period to post-reproductive life in women is called menopausal transition and is an important turning point in a woman's life cycle. Most women experience menopausal symptoms during this period and the majority of these symptoms are severe and long-lasting. Vasomotor symptoms in women can disrupt sleep, cause forgetfulness and fatigue, as well as mental changes, increase anxiety and create conditions such as depressive mood.

Non-drug methods are frequently preferred in menopausal symptoms, especially in mental effects, and their effectiveness on symptoms is remarkable. Non-drug methods mainly used in the management of postmenopausal symptoms are sports, avoiding bad habits, paying attention to diet and increasing fluid intake, wearing comfortable clothes. In addition, there are many supportive methods such as stress reduction meditation practices, garden therapies, breathing and physical exercise practices, aromatherapy. Among the most frequently used coping methods of women experiencing menopausal symptoms such as irritability and anxiety/anxiety, it was found that 'paying attention to different things (housework, cleaning, cooking, handicrafts, etc.)' was among the most frequently used coping methods. In this direction, it is thought that occupational practice may have positive effects on menopausal symptoms in women. Engagement practices are one of the methods widely used in recent years to cope with anxiety, depression and stress.

Our study aimed to measure the effectiveness of mindfulness-based practices on menopausal symptoms and psychological well-being in menopausal women by blending mindfulness-based practices and busyness practices, and in this sense, it is anticipated that it will make a significant contribution to the literature.

Objective: This study will be conducted to determine the effect of mindfulness-based and occupational practices on psychological well-being and menopausal symptoms in menopausal women.

Materials and Methods: The research will be conducted as a randomised controlled experimental study in a four-group, parallel, pretest-posttest design. The research is planned to be conducted between December 2024 and December 2025. The population of the study consists of women in menopause who applied to the ASM in the centre of Kars between December 2024 and December 2025. The sample of the study will consist of women who meet the inclusion criteria among these women. As a result of the power analysis performed in the G*Power version 3.1.9.7 programme, it was determined that a total of 76 participants, at least 19 people in each of the intervention and control groups, with a sample size, 95% confidence, 95% test power (1-ß), 0.05% margin of error level, d = 0.25 effect size (Kang, 2021). Considering 10% possible data loss in the study, it was planned to include 20 women in each of the intervention and control groups.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering to participate in the research,
* Knowing how to read and write Turkish,
* Do not be in menopause,
* Having a smart mobile phone,

Exclusion Criteria:

* Don't take hormone therapy,
* The presence of a diagnosed psychiatric illness,
* Visual, hearing, speech, physical or mental disability,
* Interruption of the application made within the scope of Engagement Practices,
* Taking psychiatric medication (antidepressants, benzodiazepines, hypnotics, narcotics, etc.), Using any other CAM method (such as Reiki, phytoestrogens, acupressure).

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-08-02 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Psychological Well-Being Scale | Eight weeks
  The scale developed by Dinner in 2009 to measure the level of psychological well-being is a 7 Likert scale consisting of 8 items. The Turkish validity and reliability of the scale was conducted in 2013. Psychological Well-being Scale defines important elements of human functioning such as positive relationships, self-efficacy perception, having a meaningful and purposeful life. The score obtained from the scale varies between 8-56. A high score indicates that the person has many psychological resources and strengths. Cronbach's alpha coefficient of the scale was found to be 0.80.
The menopause Rating Scale (MRS) | Eight weeks
  MSDS was developed by Schneider et al. in 1992. Turkish validity and reliability study was conducted in 2005. The CDSS consists of 11 items and 3 sub-dimensions. The sub-dimensions are named as 'Somatic Complaints', 'Psychological Complaints', 'Urogenital Complaints'. The scale is answered in 5-point Likert scale and each statement is scored as 0: None, 1: Mild, 2: Moderate, 3: Severe and 4: Very severe. The lowest score that can be obtained from the whole scale is 0 and the highest score is 44. An increase in the total score obtained from the scale indicates an increase in the severity of the complaints experienced and a negative impact on the quality of life. The cronbach alpha reliability coefficient of the original scale is 0.84. The cronbach alpha values of the subgroups are 0.65 for somatic complaints, 0.79 for psychological complaints and 0.72 for urogenital complaints.

CONTACTS AND LOCATIONS:
Overall Officials: Şafak Aydin, ASSISTANT PROFESSOR, Principal Investigator — Kafkas University
Locations (1):
- Kafkas University, Kars, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Telef, B.B. (2013). Psikolojik iyi oluş ölçeği: Türkçeye uyarlama, geçerlik ve güvenirlik çalışması. Hacettepe Üniversitesi Eğitim Fakültesi Dergisi, 28(28-3), 374-384.
- [Background] Gürkan, Ö.C. (2005). Menopoz semptomları değerlendirme ölçeğinin Türkçe formunun güvenirlik ve geçerliliği. Hemşirelik Forumu Dergisi, 3, 30-5.